CLINICAL TRIAL: NCT00768508
Title: Combined Pharmacotherapies for Alcoholism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bankole Johnson (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Bankole Johnson, Chair of Psychiatry and NB Sciences, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12790; R01AA012964 (NIH)
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Alcoholism
Keywords: Alcohol; Alcohol Dependence; Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Ondansetron; Cognitive Behavioral Therapy; Naltrexone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ondansetron (Experimental): Ondansetron 4 ug/kg b.i.d. + Cognitive Behavioral Therapy
  Interventions: Drug: Ondansetron 4 ug/kg b.i.d. + Cognitive Behavioral Therapy
- Naltrexone (Experimental): Naltrexone 50 mg/day + Cognitive Behavioral Therapy
  Interventions: Drug: Naltrexone 50 mg/day + Cognitive Behavioral Therapy
- Ondansetron + Naltrexone (Experimental): Ondansetron 4 ug/kg b.i.d. + Naltrexone 50 mg/day + Cognitive Behavioral Therapy
  Interventions: Drug: Ondansetron 4 ug/kg b.i.d.+ Naltrexone 50 mg/day + Cognitive Behavioral Therapy
- Placebo (Placebo Comparator): Placebo + Cognitive Behavioral Therapy
  Interventions: Other: Placebo + Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Ondansetron 4 ug/kg b.i.d. + Cognitive Behavioral Therapy — Ondansetron 4 ug/kg b.i.d.for 12 weeks
  Other Names: Zofran
  Arms: Ondansetron
Drug: Naltrexone 50 mg/day + Cognitive Behavioral Therapy — Naltrexone 50 mg/day for 12 weeks
  Other Names: Revia
  Arms: Naltrexone
Drug: Ondansetron 4 ug/kg b.i.d.+ Naltrexone 50 mg/day + Cognitive Behavioral Therapy — Combination of ondansetron 4 ug/kg b.i.d. and naltrexone 50 mg/day for 12 weeks
  Other Names: Zofran and Revia
  Arms: Ondansetron + Naltrexone
Other: Placebo + Cognitive Behavioral Therapy — Placebo comparator
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
This study would like to test whether the combination of ondansetron and naltrexone will be superior to either medication alone or placebo in the treatment of alcohol dependence.

DETAILED DESCRIPTION:
We propose to conduct a 13 week randomized, controlled clinical trial to evaluate the safety and efficacy of ondansetron and naltrexone alone and in combination.Eligible subjects will be randomized to placebo, ondansetron, naltrexone, or ondansetron + naltrexone treatments. All subjects will receive a weekly CBT (Cognitive Behavioral Therapy)sessions.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who have given written informed consent.
* Ages 18 years and above and must weigh at least 40 kg and no more than 140 kg.
* Good physical health as determined by a complete physical examination, an EKG within normal limits, and laboratory screening tests within acceptable parameters (see exclusion criteria).
* Current DSM-IV diagnosis of alcohol dependence
* AUDIT score of equal or more than 8.
* Currently drinking
* Provide evidence of stable residence in the last month prior to enrollment in the study, and have no plans to move in the next three months.
* The pregnancy test for females at intake must be negative. Additionally, women of childbearing potential must be using an acceptable form of contraception. These include: oral contraceptives, hormonal (levonorgestrel) or surgical implants, or barrier plus spermicide.
* Literate in English and able to read, understand, and complete the ratings scales and questionnaires accurately, follow instructions, and make use of the behavioral treatments.
* Answer an advertisement in the newspaper/radio/television, or be referred from a health care professional and express a wish to stop drinking.
* Willingness to participate in behavioral treatments for alcoholism.

Exclusion Criteria:

* Any current axis I DSM IV psychiatric disorder other than alcohol or nicotine dependence
* Elevation of liver enzymes - (SGOT), serum glutamic pyruvic transaminase (SGPT), blood urea nitrogen (BUN), or lactate dehydrogenase (LDH) greater than four times the normal range, or clinically significant elevated direct bilirubin as deemed by the principal investigator.
* Severe alcohol withdrawal symptoms which in the physicians opinion requires inpatient treatment.
* Serious medical co-morbidity requiring medical intervention or close supervision, or any condition which can interfere with the receipt of ondansetron.
* Severe or life-threatening adverse reactions to medications in the past or during this clinical trial.
* Female patients who are pregnant, lactating, or not adhering to an acceptable form of contraception at any time during the study.
* Received inpatient or outpatient treatment for alcohol dependence within the last 30 days (support groups such as AA are not exclusionary).
* Compelled to participate in an alcohol treatment program to maintain their liberty.
* Members of the same household.
* Concurrent treatment with any medications having a potential effect on alcohol consumption and related behaviors, or mood. These include: opiate antagonist (e.g. naltrexone), glutamate antagonists (e.g., acamprosate), serotonin re-uptake inhibitors (e.g. fluoxetine), serotonin antagonists (e.g. ritanserin or buspirone), other antidepressants (e.g. tricylic antidepressants or monoamine oxidase inhibitors), dopamine antagonists (e.g. haloperidol), calcium channel antagonists (e.g. isradipine), or compounds with actions similar to disulfiram (antabuse) or nicotine.
* Before double-blind randomization, urine must be free of opiates, cocaine, amphetamines, barbiturates, benzodiazepines, prescription and non-prescription drugs.
* Pyrexia of unknown origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2008-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Self-report measures of alcohol-related problems and consumption, Objective measures of alcohol consumption | Throughout the study
  Drinks per drinking day, Drinks per day, Percent Days Abstinent, BAC, CDT, GGT

SECONDARY OUTCOMES:
Medication compliance, alcohol craving, social functioning, quality of life, alcohol withdrawal, attendance at psychosocial services, pre-morbid risk factors | Throughout the study
  Pill Count, SFQ, AASE, ADBS, OCDS, CIWA-Ar, CGI, TCI, MAC, AOQ, FHAM

CONTACTS AND LOCATIONS:
Overall Officials: Bankole Johnson, DSc,MD,PhD, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - UVA CARE, Charlottesville, Virginia
  - UVA CARE Richmond, Richmond, Virginia